CLINICAL TRIAL: NCT01131481
Title: Evaluation of Glistenings in Intraocular Lenses AVS Model X-60 Vs AcrySof MA50-BM.
Brief Title: Evaluation of Glistenings in Intraocular Lenses Implanted in Normal Patients Following Routine Cataract Extraction.
Acronym: AVS Vs MA50BM
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Fry Eye Associates and Fry Eye Surgery Center (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Luther L. Fry,M.D., Fry Eye Associates and Fry Eye Surgery Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Protocol Number 7248
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2011-06

CONDITIONS: Glistenings
Keywords: cataracts,glistenings,intraocular lenses.
MeSH Terms: conditions — Cataract | interventions — Lenses, Intraocular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AcrySof MA50BM,AVS Model X-60 (Other): AcrySof MA50BM, AVS Model X-60
  Interventions: Device: Intraocular lens

INTERVENTIONS:
Device: Intraocular lens

SUMMARY:
Evaluation of glistenings in intraocular lenses implanted in normal patients following routine cataract surgery. The lenses used will be Model X-60 made by the AVS company Vs AcrySof MA50BM made by the Alcon company.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Bilateral cataracts requiring surgery
* Potential visual acuity of 20/40 or better in both eyes
* Require IOL power in range of 15-25 diopters
* Pupillary dilation of at least 6mm
* Willing and able to provide informed consent and attend follow-up appointments to 3 years

Exclusion Criteria:

* Any co-existing ocular disease or previous ocular surgery that would confound findings in the study, especially those effecting quality of vision. Examples include Macular degeneration amblyopia and prior epiretinal membrane peel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Glistenings between the Model X-60 made by the AVS company and AcrySof MA50BM made by the Alcon company. | The patient will be followed 1-2 days after surgery on the first eye and 1-2 days after surgery on the second eye,1-2 months after surgery on both eyes,4-6 months after surgery on both eyes and 1,2 and 3 yrs after surgery on both eyes.
  Each patient will have the same testing at each visit. Photos will be taken of the glistenings,sent off and counted.

CONTACTS AND LOCATIONS:
Overall Officials: Luther Fry, MD, Principal Investigator — Fry Eye Associates
Locations (1):
- Fry Eye Associates, Garden City, Kansas, United States